CLINICAL TRIAL: NCT00444496
Title: SPHERE Hypertension Baseline Data Study
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Hendrika Meischke, University of Washington
Other Study IDs: 06-4566-E/G 01; CDC Grant # 1 P01 CD000249-01
Record Dates: First submitted 2007-03-06; First posted 2007-03-07 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2008-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
We are collecting baseline data on patients who have high blood pressure readings (160/100 or higher) at a 9-1-1 response by an EMT.

DETAILED DESCRIPTION:
We are collecting baseline data on patients who have high blood pressure readings (160/100 or higher) at a 9-1-1 response by an EMT. We want to understand what these patients currently remember occurring during the 9-1-1 response around their high blood pressure measure; if the patients seek a second reading; if the patients seek follow-up care as a result of the high blood pressure measure. We are also interested if patients trust EMTs as a provider of preventive health care. This baseline data will also allow us to more accurately measure the success of a future intervention study aimed at motivating subjects to receive a follow-up hypertension assessment from a physician after receiving a high blood pressure reading from an EMT.

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure greater than or equal to 160 and/or diastolic blood pressure greater than or equal to 100
* Patient is at least 18 years old
* Patient was not transported by paramedics
* Patient was not admitted to a hospital
* Patient is not a nursing home/adult family home resident
* Patient's phone number is listed in the MIRF database

Exclusion Criteria:

* not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People seen by Renton, Bellevue, and Shoreline fire departments with blood pressure higher than 160/100.
Sampling Method: Probability Sample
Enrollment: 470 (Actual)
Dates: Start 2007-02; Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hendrika Meischke, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States